CLINICAL TRIAL: NCT00197158
Title: Demonstrate the Non-inferiority of Immunogenicity Elicited by GSK Biologicals' Hepatitis B Vaccine, Multidose Engerix™-B to That of Monodose Engerix™-B When Administered According to 0,1,6 Mths Schedule in Healthy Adults Aged ≥ 18 Yrs
Brief Title: Comparison of Monodose and Multidose Presentations of GSK Biologicals' Hepatitis B Vaccine in Terms of Immune Response
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 104387
Record Dates: First submitted 2005-09-15; First posted 2005-09-20 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines

INTERVENTIONS:
Biological: Hepatitis B vaccine

SUMMARY:
GSK Biologicals' currently licensed multidose hepatitis B vaccine will be compared to the currently licensed monodose hepatitis B vaccine in a population with well documented hepatitis B immunological response to the vaccine (Belgium).

DETAILED DESCRIPTION:
Randomized study with two groups. One group will receive GSK's multidose hepatitis B vaccine and the other group will receive GSK's monodose hepatitis B vaccine

ELIGIBILITY:
Inclusion criteria:

* A male or female >= 18 years of age
* Written informed consent obtained from the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* If the subject is female, she must be of non-childbearing potential, i.e. either surgically sterilized or one year post-menopausal; or, if of childbearing potential, she must be abstinent or have used adequate contraceptive precautions for 30 days prior to vaccination, have a negative pregnancy test and must agree to continue such precautions for two months after completion of the vaccination series.

Exclusion criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose. (For corticosteroids, this will mean prednisone, or equivalent, greater than or equal to 0.5 mg/kg/day. Inhaled and topical steroids are allowed.)
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 30 days of the first dose of vaccine.
* Previous vaccination against hepatitis B
* History of hepatitis B infection
* Known exposure to hepatitis B within the previous 6 weeks
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine(s).
* Acute disease at the time of enrolment. (Acute disease is defined as the presence of a moderate or severe illness with or without fever. All vaccines can be administered to persons with a minor illness such as diarrhoea, mild upper respiratory infection with or without low-grade febrile illness, i.e. Oral temperature < 37.5°C (99.5°F) / Axillary temperature <37.5°C (99.5°F).
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period. Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2005-03; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Measurement of antibody concentrations to hepatitis B antigen at Month 7.

SECONDARY OUTCOMES:
Measurement of antibody concentrations to hepatitis antigen at Months 1,2and6. Occurrence of solicited local symptoms and solicited general symptoms during the 4-day f/u period after vaccination. Occurrence, intensity and relationship to vaccination

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wilrijk, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 104387 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104387 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104387 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104387 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104387 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104387 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register